CLINICAL TRIAL: NCT01127321
Title: A Phase 1, Double-blind, Randomized, Single Ascending Dose Study of the Safety and Tolerability of MEDI-570 in SLE
Brief Title: A Safety and Tolerability Study of MEDI-570 in Systemic Lupus Erythematosus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: MedImmune LLC (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP209
Record Dates: First submitted 2010-04-14; First posted 2010-05-20 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Systemic lupus erythematosus; SLE; MEDI-570
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — MEDI-570

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): A single double-blind dose of placebo matched to MEDI-570 subcutaneous injection on Day 1.
  Interventions: Other: Placebo
- MEDI-570 0.03 MG (Experimental): A single open-label dose of MEDI-570, 0.03 milligram (mg) subcutaneous injection on Day 1.
  Interventions: Biological: MEDI-570 0.03 MG
- MEDI-570 0.1 MG (Experimental): A single open-label dose of MEDI-570, 0.1 mg subcutaneous injection on Day 1.
  Interventions: Biological: MEDI-570 0.1 MG
- MEDI-570 0.3 MG (Experimental): A single double-blind dose of MEDI-570, 0.3 mg subcutaneous injection on Day 1.
  Interventions: Biological: MEDI-570 0.3 MG
- MEDI-570 1 MG (Experimental): A single double-blind dose of MEDI-570, 1 mg subcutaneous injection on Day 1.
  Interventions: Biological: MEDI-570 1 MG

INTERVENTIONS:
Other: Placebo — A single double-blind dose of placebo matched to MEDI-570 subcutaneous injection on Day 1.
  Arms: Placebo
Biological: MEDI-570 0.03 MG — A single open-label dose of MEDI-570, 0.03 milligram (mg) subcutaneous injection on Day 1.
  Arms: MEDI-570 0.03 MG
Biological: MEDI-570 0.1 MG — A single open-label dose of MEDI-570, 0.1 mg subcutaneous injection on Day 1.
  Arms: MEDI-570 0.1 MG
Biological: MEDI-570 0.3 MG — A single double-blind dose of MEDI-570, 0.3 mg subcutaneous injection on Day 1.
  Arms: MEDI-570 0.3 MG
Biological: MEDI-570 1 MG — A single double-blind dose of MEDI-570, 1 mg subcutaneous injection on Day 1.
  Arms: MEDI-570 1 MG

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of MEDI-570 in adult subjects with moderately to severely active systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
This is a Phase 1, double-blind, randomized, placebo-controlled study to evaluate the safety and tolerability of escalating single subcutaneous doses of MEDI-570 in adult subjects with moderately to severely active SLE.

ELIGIBILITY:
Inclusion Criteria:

* Meet or have met at least 4 of the 11 revised American College of Rheumatology (ACR) classification criteria for systemic lupus erythematosus (SLE)
* Score greater than or equal to (>=) 6 points on the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) at Screening
* Ability to complete the study period, including follow-up period through Day 169
* Willingness to forego other forms of experimental treatment during the study.

Exclusion Criteria:

* History of cancer except basal cell carcinoma treated with apparent success with curative therapy >=1 year before randomization into the study
* Evidence of active or latent tuberculosis (TB)
* History of primary immunodeficiency
* Evidence of infection at any time with hepatitis B or C virus or human immunodeficiency virus (HIV)-1 or HIV-2, or active infection with hepatitis A, as determined by results of testing at Screening
* History of sepsis or serious, recurrent, chronic infection, current signs and symptoms of clinically significant chronic infection, or recent (within 6 months before Baseline visit) serious infection
* Any history or evidence of opportunistic infection within 6 months of Screening including severe cytomegalovirus (CMV) or herpetic infections (such as disseminated herpes, herpes encephalitis, ophthalmic herpes)
* Receipt of cyclophosphamide (intravenous or oral) within 6 months of Screening
* Have any absolute contraindications to skin punch biopsies, for example, a history of coagulation disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Close, PhD, Study Director — MedImmune Ltd
Locations (17):
- United States (9):
  - Research Site, Long Beach, California
  - Research Site, San Leandro, California
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Ocala, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Lansing, Michigan
  - Research Site, New York, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Columbus, Ohio
- Research Site, London, Ontario, Canada
- Mexico (3):
  - Research Site, Chihuahua City
  - Research Site, Guadalajara
  - Research Site, México
- Peru (2):
  - Research Site, Lima
  - Research Site, Trujillo
- South Africa (2):
  - Research Site, Cape Town
  - Research Site, Johannesburg

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to premature termination of the study, planned treatment cohorts, MEDI-570, 3 milligram (mg) and MEDI-570, 10 mg, were not administered. A total of 17 participants were randomized in the study. An additional 27 participants were screened but not randomized in the study.
Period: Overall Study
Arm/Group | Placebo | MEDI-570 0.03 MG | MEDI-570 0.1 MG | MEDI-570 0.3 MG | MEDI-570 1 MG
Started | 3 | 1 | 1 | 7 | 5
Completed | 3 | 1 | 1 | 7 | 5
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were randomized into the study and received at least 1 dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI-570 0.03 MG | MEDI-570 0.1 MG | MEDI-570 0.3 MG | MEDI-570 1 MG | Total
Number analyzed (Participants) | 3 | 1 | 1 | 7 | 5 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (10.6) | 49.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this group. | 41.0 (NA) — Standard deviation was not available as there was only 1 participant analyzed for this group. | 35.6 (22.2) | 39.6 (13.8) | 38.4 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 6 | 5 | 16
  Male | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received study drug. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between administration of study drug and Day 169 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Day 1 to Day 169
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Placebo | MEDI-570 0.03 MG | MEDI-570 0.1 MG | MEDI-570 0.3 MG | MEDI-570 1 MG
Number analyzed (Participants) | 3 | 1 | 1 | 7 | 5
participants
  TEAEs | 3 | 1 | 1 | 7 | 4
  TESAEs | 0 | 0 | 1 | 2 | 0

2. Secondary Outcome: Pharmacokinetic Parameters for MEDI-570
Description: Following pharmacokinetic parameters were to be evaluated by using non-compartmental analysis: t1/2 = terminal phase elimination half-life which is the time measured for the serum concentration to decrease by one half; tmax = time to maximum observed serum concentration; Cmax = maximum observed serum concentration; AUC (0-t) = area under the serum concentration-time curve from time 0 to last measurable concentration; AUC (0-infinity) = area under the serum concentration-time curve from time 0 to extrapolated infinite time obtained from AUC (0-t) plus AUC (t-infinity); Vz/F = apparent volume of distribution, which is the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug; CL/F = apparent clearance which is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: Predose and postdose on Day 1; Day 3, 5, 8, 15, 29, 57, 85, 113, 141, and 169
Population: Due to early termination of the study, the results were reported as individual participant's listings but not statistically summarized.
Arm/Group | Placebo | MEDI-570 0.03 MG | MEDI-570 0.1 MG | MEDI-570 0.3 MG | MEDI-570 1 MG
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Anti-Drug Antibodies to MEDI-570 at Any Visit
Time Frame: Predose on Day 1; Day 85, 113, and 169
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Placebo | MEDI-570 0.03 MG | MEDI-570 0.1 MG | MEDI-570 0.3 MG | MEDI-570 1 MG
Number analyzed (Participants) | 3 | 1 | 1 | 7 | 5
participants | 0 | 0 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Day 1 to Day 169
Arm/Group | Placebo | MEDI-570 0.03 MG | MEDI-570 0.1 MG | MEDI-570 0.3 MG | MEDI-570 1 MG
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1 | 1/1 | 2/7 | 0/5
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1 | 1/1 | 7/7 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=3) | MEDI-570 0.03 MG (N=1) | MEDI-570 0.1 MG (N=1) | MEDI-570 0.3 MG (N=7) | MEDI-570 1 MG (N=5)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=3) | MEDI-570 0.03 MG (N=1) | MEDI-570 0.1 MG (N=1) | MEDI-570 0.3 MG (N=7) | MEDI-570 1 MG (N=5)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
General symptom (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Administration related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cd4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vasculitic rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early by the sponsor due to business reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.